CLINICAL TRIAL: NCT07085793
Title: Prognostic Value of Estimated Plasma Volume in Patients With Acute Heart Failure
Brief Title: Estimated Plasma Volume in Patients With Acute Heart Failure
Acronym: ePVS
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: Estimated plasma volume- ePVS
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Acute Heart Failure
Keywords: Estimated plasma volume status (ePVS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: 1

SUMMARY:
Congestion plays an essential role in acute heart failure (AHF) outcomes. Estimated plasma volume status (ePVS), derived from simple hematological parameters, may offer prognostic value.

The objectif is to assess the prognostic value of admission ePVS, calculated using Duarte and Hakim formulas, for short- and long-term mortality and/or readmission in patients hospitalized for AHF.

DETAILED DESCRIPTION:
it is a prospective cross-sectional study in the emergency department of Fattouma Bourguiba University Hospital of Monastir, Tunisia.This study was approved by the Institutional Review Boardof our institute and conducted according to the revised Declaration of Helsinki. The requirement of written informed consent was waived, as this study is observational. an opt-out method was used for participant recruitment.

ePVS at admission was calculated as follows:

* Duarte ePVS= 100-ht(%) /Hb(g/dl).
* Hakim ePVS = [(actual plasma volume-ideal plasma volume)/ideal plasma volume] × 100 Actual plasma volume: (1-hematocrit) × (a+b×body weight in kg). Ideal plasma volume = c×body weight in kg. (males: a = 1530, b = 41.0, c = 39; females; a = 864, b = 47.9, c = 40)

ELIGIBILITY:
* Inclusiuon criteria :
* Patients aged over 18
* diagnosis of AHF based on clinical examination, echocardiography, the value of BNP or NT pro-BNP and expert opinion.
* Exclusion criteria :
* pregnancy
* end-stage or severe renal failure with creatinine clearance < 15 ml/min
* hemodialysis.
* refusal to consent
* Pregnant or breast feeding women.
* Alteration of consciousness GCS < 15
* Critically ill patients needing immediate mechanical hemodynamic of ventilatory support.
* Inability to follow instructions or comply with follow-up procedures.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute heart failure admetted in emergency department
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
readmission for AHF and/or all-cause mortality | 30 days
  readmission for AHF and/or all-cause mortality at 1 month
readmission for AHF and/or all-cause mortality | 365 days
  readmission for AHF and/or all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Pr, Principal Investigator — University of Monastir
Locations (1):
- Emergency Department, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No